CLINICAL TRIAL: NCT00972829
Title: Tolerability and Lipid Lowering Effect of Weekly/Biweekly Crestor in Statin Intolerant Patients Treated With Zetia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Responsible Party: Lawrence Baruch, MD, James J. Peters VA Medical Center
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: BAR-09-07
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crestor (Experimental): Crestor 10 or 20 milligrams
  Interventions: Drug: Rosuvastatin
- Ezetimibe (Active Comparator): Ezetimibe 5 or 10 milligrams
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 10 or 20 milligrams once or twice a week
  Other Names: Crestor
  Arms: Crestor
Drug: Ezetimibe — Ezetimibe 5 or 10 milligrams
  Other Names: Zetia
  Arms: Ezetimibe

SUMMARY:
Recently, research studies have shown that patients who have had trouble taking statins every day, are able to take statins if they take them only once or twice a week. The investigators are doing a research study which involves switching people who are taking ezetimibe to the statin Crestor once or twice a week and to see how ell Crestor lowers cholesterol and if it is tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of intolerance to statins
* Patients currently receiving ezetimibe
* Patients willing and able to provide signed informed consent

Exclusion Criteria:

* Patients receiving a statin (Lipitor, Crestor, Lescol, Simvastatin, or Pravachol)
* Stroke, TIA, myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass surgery, or major surgery within 3 months
* Cancer undergoing active treatment
* Creatinine clearance < 40 ml/minute
* Active liver disease or persistent elevation of SGOT or SGPT > 2 times the upper limit of normal level
* Participation in any clinical study within the last 30 days
* Drug addition or alcohol abuse within the past 6 months
* Use of cyclosporine within the last 3 months
* Use of gemfibrozil within the last month
* Patients unwilling or unable to provide informed consent
* Patients with poor compliance
* Women of childbearing potential
* History of rhabdomyolysis due to statins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-12 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Low-density lipoprotein (LDL) cholesterol | 6 weeks
Low-density lipoprotein (LDL) cholesterol | 3-4 months

SECONDARY OUTCOMES:
The ability to remain on Crestor for the study period | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Baruch, MD, Principal Investigator — James J.Peters VA Medical Center
Locations (1):
- Bronx VA Medical Center, The Bronx, New York, United States